CLINICAL TRIAL: NCT04206436
Title: CFTR Modulator Effects on Bone and Muscle in Adults With Cystic Fibrosis
Status: Active, not recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Erik Imel, Associate Professor, Indiana University
Other Study IDs: 1908566174
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis; Bone Loss; Muscle Loss
MeSH Terms: conditions — Cystic Fibrosis; Bone Diseases, Metabolic; Muscular Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples kept for batch processing at end of study. Samples may also be kept and de-identified and kept for additional testing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- on CFTR: For patients on or near time of initiation CFTR modulator therapy
  Interventions: Drug: Cftr Modulators
- Controls: controls will be patients not eligible for available treatment

INTERVENTIONS:
Drug: Cftr Modulators — CFTR modulators are drugs used to treat cystic fibrosis
  Groups: on CFTR

SUMMARY:
Study is looking at the effects of cystic fibrosis treatment on bone muscle.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a complex multisystem genetic disease, with pulmonary and gastrointestinal consequences dominating the clinical picture. The life-expectancy of CF patients has increased through several therapeutic advances. Although respiratory failure remains the major cause of mortality in CF, musculoskeletal impairments contribute to major morbidity. In the general population, musculoskeletal conditions are among the most common reasons for seeking medical care, and the risk of osteoporotic fracture increases with age. As the CF population ages, the morbidity related to musculoskeletal effects may increase.

The etiology of CF related bone disease is multifactorial and includes effects of pancreatic insufficiency, poor nutritional status, vitamin D deficiency, glucocorticoid treatment, inflammation, hypogonadism, and sarcopenia, collectively resulting in attenuated bone mineral accrual and low bone density The effect of cystic fibrosis transmembrane conductance regulator (CFTR) modulating drugs on bone disease in CF has not been evaluated. Effects of CFTR modulators may help counter the bone and muscle consequences of CF either directly by effects on bone or muscle cells, or indirectly by improved lung disease, improved nutritional status, decreased systemic inflammation or glucocorticoid use, or subsequent increases in physical activity.

The rationale that underlies the proposed research is that better understanding of the bone and muscle effects of CFTR modulator therapies will help guide strategies to optimize bone accrual, prevent osteoporosis and fractures, and improve functional outcomes in the aging CF population. Set on the backbone of a longitudinal observational cohort study, the study will systematically and comprehensively evaluate changes in bone and muscle mass and strength from baseline to 12 month and 24 month time points among patients receiving CFTR modulator therapies and also among controls not receiving CFTR modulator therapies.

ELIGIBILITY:
Inclusion Criteria:

* documented, confirmed diagnosis of CF

  * Age ≥18 years old
  * >21 days since the start of their last pulmonary exacerbation at the baseline visit
  * Provide signed written informed consent to participate

Exclusion Criteria:

* • Estimated glomerular filtration rate (eGFR) <30 ml/min/m2 using the CKD-EPI equation,

  * Treatment with any osteoporosis medication within 6 months for oral agents or 1 year for intravenous or injectable agents (Subjects may participate if therapy stopped earlier than these time periods).
  * Current treatment with growth hormone or IGF-1
  * Currently pregnant or lactating or planning plan on becoming pregnant during the duration of the study.
  * Life expectancy less than 12 months
  * History of lung transplantation
  * Conditions that in the opinion of the investigators would interfere with the ability to collect or interpret the data, or put the patient at higher safety risk from study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment will target groups that are frequency matched for age (decade), race, sex, pancreatic insufficiency and glucocorticoid usage (inhaled or systemic as both have skeletal effects in some studies) to control for these factors influencing relevant bone and muscle outcomes. (see statistical description). The study will enroll up to 30 subjects in each group, expecting up to 25% dropout.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify the effects of CFTR modulators on bone mineral density | 12 months
  Changes from baseline to 12 month in total volumetric BMD and in estimated failure load as measured by HRpQCT at the distal radius and tibia
establish the effect of CFTR modulators on sarcopenia. | 12 months
  changes from baseline to 12 months in whole body lean mass using body composition software on DXA

SECONDARY OUTCOMES:
Identify the effect of CFTR modulators on bone mineral density | 6, 12 and 24 month
  Changes from baseline to 24 month in total volumetric BMD and in estimated failure load as measured by HRpQCT at the distal radius and tibia.
  Changes from baseline to 6, 12, and 24 month in HRpQCT measure of cortical vBMD and trabecular vBMD at both the distal radius and tibia and cortical vBMD and trabecular vBMD at diaphyseal site.
  Changes from baseline to 6, 12 and 24 month in HRpQCT measure of cortical vBMC and trabecular vBMD at both the distal radius and tibia and cortical vBMD at a diaphyseal site Changes from baseline to 6,12, and 24 month in areal BMD using DXA at eh lumbar spine, total body, femur neck and total hip
establish the effect of CFTR modulators on sarcopenia. | 6, 12 and 24 month
  changes from baseline to 6 and 24 months in whole body lean mass using body composition software on DXA Changes from baseline to 6, 12, 24 months in appendicular lean mass relative to height measured using body composition software on DXA

CONTACTS AND LOCATIONS:
Overall Officials: Erik A Imel, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No